CLINICAL TRIAL: NCT03520595
Title: Analgesic Efficacy of Arnica Montana in Comparison With Diclofenac Sodium Following a Periodontal Surgical Procedure: A Placebo Control Trial
Brief Title: Analgesic Efficacy of Arnica Montana in Comparison With Diclofenac Sodium Following a Periodontal Surgical Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr.Nibha Suneel Kulkarni, Principal Investigator, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tatyasaheb kore dental c
Record Dates: First submitted 2017-01-31; First posted 2018-05-11 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Crown Lengthening Procedure With Ostectomy
MeSH Terms: interventions — cysteine and glycine-rich protein 3; Diclofenac

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Arnica Group (Active Comparator): Study group 1 CLP with ostectomy Arnica 200 drug 3 pills,3 times daily for 3 days
  Interventions: Drug: Arnica 200 drug 3 pills,3 times daily for 3 days
- Diclofenac Sodium group (Active Comparator): Study group 2 CLP with ostectomy Diclofenac Sodium 50mg twice daily after meals with plain water
  Interventions: Drug: Diclofenac Sodium 50mg twice daily
- Placebo Group (Placebo Comparator): Study group 3 CLP with ostectomy Placebo pills and distilled water 3 pills,3 times daily
  Interventions: Drug: Placebo pills and distilled water 3 pills,3 times daily

INTERVENTIONS:
Drug: Arnica 200 drug 3 pills,3 times daily for 3 days — CLP with ostectomy done in patients whose biologic width and crown height is insufficient
  Other Names: CLP with ostectomy
  Arms: Arnica Group
Drug: Diclofenac Sodium 50mg twice daily — CLP with ostectomy done in patients whose biologic width and crown height is insufficient
  Other Names: CLP with ostectomy
  Arms: Diclofenac Sodium group
Drug: Placebo pills and distilled water 3 pills,3 times daily — CLP with ostectomy done in patients whose biologic width and crown height is insufficient
  Other Names: CLP with ostectomy
  Arms: Placebo Group

SUMMARY:
Introduction:

Homeopathy is a deep healing, comprehensive and distinct system originally developed by Samuel Hahnemann about 200 years ago. Small doses of specially prepared ("potentized") remedies which set the body's systems back in order and stimulate a body's own energies toward a natural healing process. It is entirely distinct in both theory and in practice from other healing systems from ordinary or main-stream ("allopathic") medicine, but also from acupuncture, naturopathy, chiropractics, etc., although some homeopathy often finds its way into these other fields of practice.Homeopathy is based on the concept "similia similibus curentur" which means symptoms, caused by the original substance in healthy subjects, can be reversed by the homeopathic remedy in patients having similar symptoms.Homeopathy has the advantages such as it is inexpensive (the only expense is the homeopath's time and training - the remedies themselves cost practically nothing), non-toxic (although "side affects" which reflect the body's own healing processes may occur - such as fever, discharge, rash, etc.) and non-intrusive (the remedies are carried on tiny sugar granules which are dissolved in water or in the mouth, or swallowed).Arnica is one of the most popular medications in homeopathy medicine. This remedy can be extracted from several plant species belonging to the Aesteraceae family including Arnica montana, Arnica fulgens, Arnica cordifolia, Arnica chamissonis and Arnica sororia, and it is widely sold as tincture, ointment, cream, gel, and tablet. It has been used for the treatment of numerous pathological conditions, including pain, swelling and stiffness associated with trauma, contusions, sprains, myocarditis, angina pectoris, cardiac insufficiency, arteriosclerosis, postoperative clinical conditions, and for symptomatic relief in osteoarthritis.Conventional NSAIDs work by inhibiting cyclooxygenase (COX) and prostaglandin synthesis as well as by other less understood mechanisms. Onset of analgesia occurs rapidly with all NSAIDs, usually within one hour.Diclofenac is one of potent, standard and most unique NSAID for the therapy of postoperative pain. Diclofenac inhibits the lipoxygenase pathways, which reduces the formation of the leukotrienes (also pro-inflammatory autacoids) and also inhibit phospholipase A2. These actions explain the high potency of diclofenac.NSAIDs cause a variety of side effects including nausea, diarrhea, constipation, dizziness, headache, confusion, edema, rash, and pruritis. They can also cause more serious toxicities such as gastrointestinal (GI) ulceration/bleeding, hematologic disturbances, bronchospasm, angioedema, renal dysfunction, and hepatotoxicity. Many of these side effects are due to NSAID inhibiting prostaglandin synthesis other than at the desired site of action.Arnica being clinical efficient and high tolerable makes it a potential therapeutic alternative target to non-steroidal anti-inflammatory drugs.In this study investigator will compare and evaluate the efficacy of Arnica as a substitute for analgesics such as Diclofenac Sodium, through which side effects of NSAIDS can be avoided and get the same analgesia effect through Arnica without any of the undesirable effects for minor surgical procedures.

AIM:

To compare and evaluate the analgesic effect of Arnica Montana with Diclofenac sodium after crown lengthening procedure with ostectomy.

Objectives:

To assess the analgesic effect on crown lengthening procedure with ostectomy patients of Arnica Montana and Diclofenac Sodium.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients.
* Patients with inadequate crown height for replacement for prosthesis.

Exclusion Criteria:

* Tobacco intake in any form and alcohol.
* Pregnant & lactating women.
* Any known/reported allergy to given drugs.
* On Antibiotics medications.
* Patient with the history of acidity ,gastric disorders.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 3 days
  Pain Assessment is done by visual analog scale which consists of 10 centimeter line. anchored by two extremes starting from 1 ending to 10, of which 1 being the lowest and 10 being highest score.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental, Kolhāpur, Maharashtra, India